CLINICAL TRIAL: NCT07272083
Title: Application of the New Diagnostic Criteria CEUS (Contrast-Enhanced Ultrasound) LI-RADS (Liver Imaging Reporting and Data System) TRA (Nonradiation Treatment Response Assessment) in the Evaluation Response to Ablation Treatment (Radiofrequency or Microwave Ablation) of Hepatocellular Carcinoma (HCC) Nodules.
Brief Title: New Diagnostic Criteria in the Evaluation Response to Ablation Treatment of Hepatocellular Carcinoma Nodules
Acronym: CEUS_LR_TRA
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 8154
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Contrast-Enhanced Ultrasound — Application of the newly updated LI-RADS CEUS Non-Radiation TRA v2024 criteria in patients undergoing ultrasound-guided locoregional thermal ablation for HCC.

SUMMARY:
Hepatocellular carcinoma (HCC) is a primary liver malignancy that typically develops in the setting of chronic liver disease with a cirrhotic background. Currently, one of the main imaging techniques used to evaluate space-occupying lesions in the splanchnic district is contrast-enhanced ultrasound (CEUS), which is characterized by high sensitivity and specificity in lesion characterization through the assessment of enhancement patterns following contrast administration.

When an HCC nodule is small (<3 cm), hepatic function is preserved, and no extrahepatic disease is present, locoregional ultrasound-guided thermal ablation-either radiofrequency ablation (RFA) or microwave ablation (MWA)-is indicated as a treatment option. In 2024, the CEUS LI-RADS (Contrast-Enhanced Ultrasound Liver Imaging Reporting and Data System) criteria were further expanded to include the Non-Radiation Treatment Response Assessment (TRA). This represents a diagnostic algorithm applied to CEUS images to provide a standardized classification of treatment response following locoregional therapies or surgical resection of hepatic malignancies (HCC, intrahepatic cholangiocarcinoma, or mixed tumors) in patients at high risk for HCC. The algorithm focuses on evaluating the characteristics of any viable tumor remnants within or immediately adjacent to a treated lesion.

The primary objective of this study is to assess the diagnostic accuracy of the newly updated LI-RADS CEUS Non-Radiation TRA v2024 criteria in patients undergoing ultrasound-guided locoregional thermal ablation for HCC.

This prospective, observational, single-center study will enroll adult patients with a diagnosis of HCC who undergo RFA or MWA at our institution. Study results will be analyzed to determine the sensitivity, specificity, area under the curve (AUC), positive predictive value (PPV), and negative predictive value (NPV) of the CEUS LI-RADS Non-Radiation TRA criteria for the rule-in and rule-out of disease recurrence.

The findings have the potential to improve patient prognosis and optimize clinical management strategies by reducing the use of second-level imaging modalities that involve ionizing radiation or nephrotoxic contrast agents.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years;
* HCC nodules treated with locoregional thermal ablation using RFA or MWA;
* Signed informed consent.

Exclusion Criteria:

* Refusal to participate in the study;
* Contraindications to performing post-treatment CEUS;
* Absence of at least one CEUS examination during follow-up after locoregional thermal ablation with RFA or MWA;
* Contraindications to performing post-treatment CT or MRI.
* Absence of post-treatment CT or MRI follow-up imaging;
* LR-TRA Nonevaluable categorization on post-treatment CT or MRI follow-up imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Enrolled patients will be adults of both sexes with a diagnosis of HCC and an indication for locoregional thermal ablation with RFA or MWA, referred to the Diagnostic and Interventional Ultrasound Unit. As per clinical practice, after locoregional treatment and when the treated lesion is visible on B-mode imaging, patients will undergo CEUS approximately 24-48 hours after the procedure (early CEUS) and subsequently at about 4 weeks with CEUS (late CEUS) and MRI/CT
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Concordance between CEUS LR-TRA and MRI/CT LR-TRA | 3 months after ablation
  Determining the concordance between CEUS LR-TRA and MRI/CT LR-TRA, by assessing the agreement between the two diagnostic techniques through the analysis of categorical variables.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Riccardi, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Università Cattolica del Sacro Cuore, Fondazione Policlinico Universitario Gemelli IRCCS, Roma, Italia, Roma, Italy

IPD SHARING:
Plan to Share IPD: No